CLINICAL TRIAL: NCT05161585
Title: Evaluation of Circulating Tumor DNA Guided Surveillance Strategy of Stage III Colorectal Cancer: an Open, Prospective, Randomized Controlled Cohort Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junjie Peng, Department of Colorectal Surgery，Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ctDNA- phaseIIICRC
Record Dates: First submitted 2021-11-21; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Stage III Colorectal Cancer; Circulating Tumor DNA
Keywords: Surveillance strategy; Stage III colorectal cancer; Circulating tumor DNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Masking Description: Postoperative adjuvant therapy (chemotherapy and radiotherapy) and specific implementation scheme shall be determined by the clinical physician blinded to ctDNA status and randomized group. Other parts are open-label.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA dynamic monitoring + routine postoperative follow-up (Experimental): ctDNA is detected before operation, before chemotherapy, and then every three months for 2 years, 10 times in total. At the same time, routine postoperative follow-up is given.
  To be pointed out, after the completion of the adjuvant chemotherapy, if the ctDNA test indicates positive, patients will immediately perform chest, abdominal and pelvic CT and other imaging tests to determine whether there is recurrence /metastasis. If it is not confirmed, repeat the imaging review every two months, and continue to perform ctDNA test every three months. If the following ctDNA test is negative for two consecutive times, the above imaging reexamination will return to the routine follow-up frequency. In addition, during the follow-up, the following situations may occur: the imaging examination has found recurrence/metastasis, but the ctDNA test is still negative. At this time, the patient will be informed and treated in time of the recurrence/metastasis.
  Interventions: Diagnostic Test: ctDNA dynamic monitoring
- routine postoperative follow-up (No Intervention): Only routine postoperative follow-up is given as follows: Physical examination and CEA were performed every 3-6 months for the first 2 years, every 6 months within the third to fifth year, and then annually. Chest/abdominal/pelvis computed tomography was performed annually for up to 5 years, and colonoscopy was performed for proper patients the first year after treatment and repeated in the third year if no advanced adenoma was found and then every 5 years.

INTERVENTIONS:
Diagnostic Test: ctDNA dynamic monitoring — ctDNA is detected before operation, before chemotherapy, and then every three months for 2 years, 10 times in total.
  Arms: ctDNA dynamic monitoring + routine postoperative follow-up

SUMMARY:
For patients with stage III colon cancers, radical resection of primary tumor followed by adjuvant chemotherapy is currently the standard treatment. Adjuvant chemotherapy with 5-fluorouracil and oxaliplatin based regimen has been proved effective to improve recurrence-free survival and overall survival. Approximately half of patients with stage III colon cancers can be cured by surgery alone, while a substantial number of patients still experience recurrence, even with standard adjuvant chemotherapy. In recent years, circulating tumor DNA (ctDNA) has been detected in the cell-free component of peripheral blood samples in advanced colorectal cancers and many other solid tumors. Several previous studies have suggested that in patients with stage I-III colorectal cancer, postoperative ctDNA was an valuable biomarker to predict minimal residual disease (MRD) after radical resection, thus redefining patients risk outcome groups and guiding postoperative treatment. In addition, recent studies based on serial postoperative ctDNA detection showed that serial ctDNA analyses revealed disease recurrence up to 5-16.5 months ahead of radiological imaging. Here, based on the role of ctDNA in predicting MRD, we conducted an open, prospective, randomized controlled phase II cohort study to explore if ctDNA can as a biomarker to guide personalized surveillance strategy after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤80 years old, regardless of gender;
* Personal status (PS) score as over 80 or Eastern Cooperative Oncology Group (ECOG) score as 0 ~ 2;
* Pathologically confirmed as stage III colorectal cancer;
* Radical operation performed ;
* With expected survival of more than 12 months;
* The subjects (or their legal representative / Guardian) must sign the informed consent form, indicating that they understand the purpose of the study, understand the necessary procedures of the study, and are willing to participate in the study.

Exclusion Criteria:

* Neoadjuvant therapy performed before operation;
* Blood transfusion performed during operation or within 2 weeks before operation;
* Incomplete baseline samples, including preoperative plasma samples, surgical tumor tissue samples and plasma samples 3-7 days after operation;
* Two consecutive test points missing or three plasma samples missing in total before a positive ctDNA time point
* Pregnant or lactating women who have fertility and do not take adequate contraceptive measures;
* Have a history of other malignant tumors within 5 years, except cured cervical carcinoma in situ or non melanoma skin cancer;
* Primary brain tumor or central nerve metastasis is not under control, with obvious intracranial hypertension or neuropsychiatric symptoms;
* Patients with the following serious or uncontrollable diseases: severe heart disease, the condition is still unstable after treatment, including myocardial infarction, congestive heart failure, unstable angina pectoris, pericardial effusion with obvious symptoms or unstable arrhythmia within 6 months before enrollment; definite neuropathy or psychosis, including dementia or seizures; severe or uncontrolled infection; active disseminated intravascular coagulation and obvious bleeding tendency;
* Significant impairment of important organ function;
* Other conditions in which the investigator believes that the patient should not participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of postoperative ctDNA in monitoring recurrence and metastasis | Up to 60 months.
  Number of patients with ctDNA positive and imaging confirmed recurrence or metastasis / number of all imaging confirmed recurrence or metastasis
Specificity of postoperative ctDNA in monitoring recurrence and metastasis | Up to 60 months.
  Number of patients with ctDNA negative and no recurrence and metastasis confirmed by imaging / number of patients with no recurrence and metastasis confirmed by imaging
Accuracy of postoperative ctDNA in monitoring recurrence and metastasis | Up to 60 months.
  True positive+True negative/sample size
Secondary resection rate | Up to 60 months.
  The rate of R0 resection for recurrence or metastasis after surgery of the primary

SECONDARY OUTCOMES:
ctDNA-disease free survival (DFS) | Under ctDNA monitoring, from date of randomization until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months.
  Disease free survival time under ctDNA monitoring
CT-DFS | Under imaging monitoring, from date of randomization until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months.
  Disease free survival time under imaging monitoring
△DFS | Up to 60 months.
  The difference between ctDNA-DFS and CT-DFS
overall survival (OS) | From date of randomization until the date of first documented date of death from any cause, assessed up to 60 months.
  Overall survival of included patients
ctDNA clearance rate | Up to 60 months.
  The rate of ctDNA positive before chemotherapy that turns negative after adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China